CLINICAL TRIAL: NCT00814333
Title: A Randomized Controlled Trial Comparing Outcomes in Patients Treated With Merocel Packing or Thrombin-JMI for Anterior Epistaxis
Brief Title: Trial Comparing Outcomes With Merocel Packing or Thrombin-JMI for Anterior Epistaxis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product supplier change - bought out. Unable to enroll patients.
Sponsor: University of Kansas Medical Center (Other)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Keith Sale, MD, Associate Professor & Vice Chairman, Otolaryngology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11564
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Epistaxis
Keywords: epistaxis
MeSH Terms: conditions — Epistaxis | interventions — Thrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Thrombin-JMI
  Interventions: Drug: Thrombin-JMI
- 2 (Active Comparator): Merocel pack
  Interventions: Drug: Merocel pack

INTERVENTIONS:
Drug: Thrombin-JMI — 5,000 IU, to nasal mucosa via syringe spray applicator
  Arms: 1
Drug: Merocel pack — 8 cm pack, inserted within the affected side between the septum and inferior turbinate via bayonet forceps
  Arms: 2

SUMMARY:
Epistaxis is a common problem among people of all ages and backgrounds. However, occasionally epistaxis can be severe enough to require emergency room admission. Among the treatment options for epistaxis, nasal packing is the most common approach. This approach requires a return visit to the clinic for removal of the packing. Additionally, there is a great deal of pain during the insertion and removal of this packing. This study aims to justify the further investigation of thrombin as a potential treatment approach for these patients. Thrombin could provide a treatment approach that reduces pain and eliminates the need for a return visit to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults that have failed first line therapy for anterior epistaxis in the ER or the hospital

Exclusion Criteria:

* Non-english speaking patients
* Patients with bleeding disorders
* Known pregnant women or women that think they may be pregnant
* Patients with a know presence of antibodies to bovine thrombin preparations
* Patients that currently have or are known to have a history of systemic skin condition or rash such as eczema or psoriasis
* Patients found to have posterior epistaxis
* Patients requiring a surrogate for medical decisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sale, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Merocel Pack: Standard of care for persons being treated for epistaxis.
  Merocel pack: 8 cm pack, inserted within the affected side between the septum and inferior turbinate via bayonet forceps
Period: Enrollment
Arm/Group | Merocel Pack | Thrombin-JMI
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Treatment Period
Arm/Group | Merocel Pack | Thrombin-JMI
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Merocel Pack | Thrombin-JMI | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Cessation of Epistaxis
Time Frame: baseline, day 4-6
Population: No participants started treatment on this study. Study was closed before any study related procedures were administered.
Arm/Group | Merocel Pack | Thrombin-JMI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Merocel Pack | Thrombin-JMI
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes